CLINICAL TRIAL: NCT02453425
Title: Goal Directed Therapy in Septic Shock - the Effects of Mean Arterial Pressure Levels, Adjusted With Norepinephrine, on Renal Perfusion, Function and Oxygenation.
Brief Title: The Effects of Blood Pressure on Renal Function and Oxygenation in Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jenny Skytte Larsson, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Sepsis-studien
Record Dates: First submitted 2015-04-23; First posted 2015-05-25 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Septic Shock; Acute Kidney Injury
Keywords: renal blood flow; renal oxygenation; glomerular filtration rate; filtration fraction; blood pressure
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 60 mmHg (Active Comparator): Norepinephrine adjusted to reach MAP 60 mmHg
  Interventions: Other: MAP 60 mmHg
- 75 mmHg (Active Comparator): Norepinephrine adjusted to reach MAP 75 mmHg
  Interventions: Other: MAP 75 mmHg
- 90 mmHg (Active Comparator): Norepinephrine adjusted to reach MAP 90 mmHg
  Interventions: Other: MAP 90 mmHg

INTERVENTIONS:
Other: MAP 60 mmHg — Norepinephrine adjusted to reach MAP 60 mmHg
  Other Names: Norepinephrine
  Arms: 60 mmHg
Other: MAP 75 mmHg — Norepinephrine adjusted to reach MAP 75 mmHg
  Other Names: Norepinephrine
  Arms: 75 mmHg
Other: MAP 90 mmHg — Norepinephrine adjusted to reach MAP 90 mmHg
  Other Names: Norepinephrine
  Arms: 90 mmHg

SUMMARY:
The purpose of this study is to evaluate renal effects of 3 different levels of mean arterial pressure in early case of septic shock. In 8 patients diagnosed with early septic shock, we will adjust mean arterial pressure (MAP) to three different levels, using norepinephrine. At each level of MAP, central and renal hemodynamics and oxygenation states will be measured. Analysis will be made to describe the pathophysiology at MAP 75 mmHg, and then to evaluate at which MAP renal function and oxygenation is least affected negatively.

DETAILED DESCRIPTION:
It is under debate what level of mean arterial pressure is the most appropriate for organ perfusion in septic shock. The kidneys are usually used for end-organ evaluation of appropriate perfusion and appropriate blood pressure level. What "adequate blood pressure" means is today unclear.

The purpose of this study is to chart the renal perfusion, oxygenation and function, and moreover to evaluate renal effects of 3 different levels of mean arterial pressure, in early phase of septic shock.

Patients will be included within the first 24 hrs after admission to the ICU diagnosed with septic shock. The patients will be sedated, mechanically ventilated and in need for norepinephrine for adequate blood pressure levels.

After 60 mins of steady state at MAP 75 mmHg, norepinephrine will be adjusted achieve MAP of 60 and 90 mmHg respectively, MAP being held at each level for 30 mins. At the end of each 30 mins period, central and renal hemodynamics will be measured, blood and urine samples will be collected.

Central hemodynamics will be measured by, and blood samples collected via a pulmonary catheter and an arterial line.

Renal hemodynamics will be measured using a renal vein catheter for retrograde thermodilution giving at hand renal blood flow (RBF), renal vein blood samples and urine collection provides extraction of Cr-EDTA for filtration fraction (FF) and glomerular filtration rate (GFR), renal oxygen consumption, and renal oxygen extraction as a measure of balance between renal oxygen delivery and consumption.

Via renal vein catheterisation and retrograde thermodilution, the study group have the unique possibility to actually evaluate renal blood flow, renal oxygenation and renal function in humans in vivo.

After finishing the data collection, analysis will be made to answer the question: which MAP is the most optimal concerning RBF, GFR and renal oxygenation in patients with septic shock?

ELIGIBILITY:
Inclusion Criteria:

* stable septic shock
* normovolemic
* norepinephrine
* intubated/ventilated
* normal s-creatinine according to local laboratory regards.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) | 195 min
  Renal function, ml/min

SECONDARY OUTCOMES:
Renal Blood Flow (RBF) | 195 mins
  ml/min
Renal Oxygen consumption | 195 mins
  ml/min
Filtration fraction | 195 mins
  glomerular filtration rate (GFR) to the renal plasma flow (RPF). Filtration Fraction, Ratio of GFR to renal plasma flow, %
Renal oxygen supply/demand relationship | 195 min
  Renal oxygen consumption compared to renal oxygen delivery (CaO2-CrvO2/CaO2).

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Professor, Study Chair — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, dpt of anesthesiology and intensive care, Gothenburg, VGR, Sweden